CLINICAL TRIAL: NCT01432210
Title: Enhancing Human Intestinal Absorption of Carotenoids and Bioconversion of Carotene to Vitamin A in the Presence of Hass Avocados
Brief Title: Provitamin A Absorption and Conversion With Avocados
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Hass Avocado Board (Other)
Responsible Party: Principal Investigator, Jessica Cooperstone, Research Scientist, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2011H0159; 60030575 (Other: OSURF)
Record Dates: First submitted 2011-09-04; First posted 2011-09-12 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: post-prandial absorption; provitamin A carotenoids; vitamin A; avocado; tomato; carrot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tomato Meal (Other): A tomato meal will be fed with and without avocado.
  Interventions: Other: Post-prandial Feeding Study
- Carrot Meal (Other): A carrot meal will be fed with and without avocado.
  Interventions: Other: Post-prandial Feeding Study

INTERVENTIONS:
Other: Post-prandial Feeding Study

SUMMARY:
Vitamin A is necessary in the human diet. The form of vitamin A found in fruits and vegetables is not "active" and must be converted to the active form in the human body. However, information on the ability of humans to absorb and convert vitamin A to the active form is still lacking. In this study, the investigators will observe the absorption and conversion of vitamin A from orange tomato sauce and/or carrots after a meal with fat (from avocado fruit) and a meal without fat. The investigators will also test whether eating these foods might protect the blood against damage that could lead to heart disease.

DETAILED DESCRIPTION:
The primary objective of this study will be to demonstrate that adding avocados to a carotene rich meal will promote the absorption of provitamin A carotenoids and enhance the delivery of greater quantities of vitamin A. This objective will be accomplished by quantitation of the immediate post-prandial plasma concentrations of parent carotenoids and vitamin A metabolites after subjects consume a meal with or without avocado in combination with a serving of tomato sauce (containing nutritionally relevant amounts of beta-carotene) or carrots.

The secondary objective of this study will be to determine if higher levels of carotenoids and other antioxidants transported in the bloodstream will have a protective role in promoting cardiovascular health. This objective will be accomplished by testing the oxidation capacity of lipoprotein fractions before and after meal supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Total cholesterol (140 to 200 mg/dL)
* BMI 17 to 30
* Age 18-70 years

Exclusion Criteria:

* Lactating, pregnant, or plan to be pregnant during study
* Tobacco use (cigarettes or chewing tobacco)
* Metabolic disease
* Malabsorption disorders
* History of cancer, esophageal, gastric, or intestinal ulcers
* History of liver or kidney insufficiency or failure
* Allergies to tomatoes or tomato products
* Allergies to carrots
* Allergies to avocados
* Obesity (BMI>30)
* Hypercholesterolemia (total cholesterol> 200mg/dL)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Post-prandial levels of provitamin A and vitamin A | Nine post-prandial blood samples will be taken over twelve hours
  The absorption of and conversion of provitamin A carotenoids into vitamin A will be measured after the consumption of a carotenoid-rich meal. The meal will be served both with and without avocado as a source of lipid.

SECONDARY OUTCOMES:
post-prandial antioxidant status of blood | comparing baseline vs. 5 hour status
  The ability of a carotenoid-rich meal to reduce the susceptibility of blood lipoproteins to oxidative stress will be tested. A modified trolox equivalent antioxidant capacity (TEAC) assay will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Schwartz, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Clinical Research Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Cooperstone JL, Goetz HJ, Riedl KM, Harrison EH, Schwartz SJ, Kopec RE. Relative contribution of alpha-carotene to postprandial vitamin A concentrations in healthy humans after carrot consumption. Am J Clin Nutr. 2017 Jul;106(1):59-66. doi: 10.3945/ajcn.116.150821. Epub 2017 May 17. PMID 28515067
- [Derived] Kopec RE, Cooperstone JL, Schweiggert RM, Young GS, Harrison EH, Francis DM, Clinton SK, Schwartz SJ. Avocado consumption enhances human postprandial provitamin A absorption and conversion from a novel high-beta-carotene tomato sauce and from carrots. J Nutr. 2014 Aug;144(8):1158-66. doi: 10.3945/jn.113.187674. Epub 2014 Jun 4. PMID 24899156